CLINICAL TRIAL: NCT06594120
Title: Veränderungen Der Arbeitsfähigkeit Und Erwerbstätigkeit Infolge Des Medizinisch Berufsorientierten Rehabilitationsverfahrens PV RehaJET [Changes in Workability and Employment Following the Work-related Medical Rehabilitation PV RehaJET]
Brief Title: Changes in Workability and Employment Following the Work-related Medical Rehabilitation PV RehaJET
Status: Recruiting | Type: Observational
Sponsor: Pensionsversicherungsanstalt (Other)
Responsible Party: Sponsor
Other Study IDs: 0031 Studie PVRehaJET als EV
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2024-09

CONDITIONS: Musculoskeletal Diseases or Conditions
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- 3-week work-specific rehabilitation: This group is referred to the work-specific rehabilitation programme immediately upon arrival at the rehabilitation centre.
  Interventions: Behavioral: Multimodal rehabilitation with additional work specific training
- 4-week work-specific rehabilitation: This group first underwent a three-week medical-focused rehabilitation programme prior to commencing the work-specific rehabilitation programme.
  Interventions: Behavioral: Multimodal rehabilitation with additional work specific training

INTERVENTIONS:
Behavioral: Multimodal rehabilitation with additional work specific training — The rehabilitation is based on the biopsychosocial ICF model of the WHO. Taking into account the physical and psychological condition of the patients, an individual therapy plan is created that is tailored to the needs of the patients.

SUMMARY:
The objective of this observational study is to gain insight into a new approach to rehabilitation in Austria, with a particular focus on work-specific exercises that are dependent on the specific work-related needs of the patients. Two groups are being observed: one was referred to a three-week work-specific rehabilitation programme immediately upon arrival at the rehabilitation centre, while the other group underwent a three-week medical-focused rehabilitation programme before starting a four-week work-specific rehabilitation programme.

Researchers will monitor for indications of improvement following completion of the rehabilitation program. As the two forms of rehabilitation are not directly comparable, they will be observed and analysed as two distinct entities.

As part of their regular inpatient rehabilitation, participants will complete questionnaires at designated intervals (beginning and end of stay), with follow-up assessments scheduled at six and 12 months post-rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* The study participants are regular patients in the rehabilitation centre Bad Hofgastein
* Presence of a disease in the area of the musculoskeletal system
* Sufficient motivation to maintain professional participation
* Declaration of consent

Exclusion Criteria:

* No completion of all work-specific rehabilitation modules
* Acute or decompensated disease states with severe functional limitations (i.e. not able to continue with the rehabilitation programme)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with specific work-related rehabilitation needs
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-08-22 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
IMBA - Profile comparison | 3 or 4 weeks of inpatient rehabilitation
  IMBA is a profile comparison method for prevention and rehabilitation. Job requirements and human capabilities are described by standardised, defined characteristics and compared directly with each other. The respective profile sheets consist, among other things, of 70 function-, activity- and context-related main characteristics in which the extent of excessive demands for each characteristic is documented on a scale of 0 - 6 (Min. = 0, Max = 420). Lower values indicate less excessive demands.
Employment history | 6 and 12 months after finishing rehabilitation
  The existence of gainful employment subject to social insurance contributions in a specific period allows conclusions to be drawn about the employment history of the rehabilitants.

SECONDARY OUTCOMES:
Work ability index (WAI) | 3 or 4 weeks of inpatient rehabilitation + 6 and 12 months after finishing rehabilitation
  The Work Ability Index (WAI) is an instrument for assessing work ability. (Min. = 7, Max = 49). Lower values indicate less subjective work ability.
Patient Health Questionnaire-4 (PHQ-4) | 3 or 4 weeks of inpatient rehabilitation + 6 and 12 months after finishing rehabilitation
  The Patient Health Questionnaire-4 (PHQ-4) operationalizes core criteria for anxiety and depression on a 4 point likert scale (Min. = 0, Max = 4). Lower values indicate less impairments.
European Quality of Life 5 Dimensions 5 Level (EQ-5D-5L) | 3 or 4 weeks of inpatient rehabilitation + 6 and 12 months after finishing rehabilitation
  The EQ-5D-5L is a general instrument for measuring patient-reported outcomes (PROs), which can be used to assess the quality of life of patients on different dimensions (mobility, self-care, usual activities, pain/discomfort) on a 5-level scale (Min. = 0, Max. = 5). Lower values indicate less impairments in the respective dimensions.
  Moreover, the EQ-5D-5L assesses the patient's self-rated health on a 100 point visual analog scale (Min. = 0, Max. = 100). Lower values indicate less positive ratings of health.

CONTACTS AND LOCATIONS:
Overall Officials: Doreen Stöhr, Mag., Study Chair — Pensionsversicherungsanstalt
Locations (1):
- Rehabilitationszentrum Bad Hofgastein, Bad Hofgastein, Salzburg, Austria